CLINICAL TRIAL: NCT00609531
Title: Functional MRI Evaluation of the Effect of Citalopram in Autism Spectrum Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gabriel Dichter, Associate Professor of Psychiatry, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 04-0975; NIH/NCRR K12 RR023248; The Dana Foundation; K23MH081285 (NIH)
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Autism Spectrum Disorders
Keywords: Restricted repetitive behaviors; restricted interests; Aspergers; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Individuals with an Autism Spectrum Disorder receiving citalopram
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Individuals with an Autistic Spectrum Disorder receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — Pill, 5-20mg once a day for twelve weeks
  Other Names: Celexa
  Arms: Active
Drug: Placebo — Placebo pill once a day for twelve weeks
  Arms: Placebo

SUMMARY:
The purpose of this proof of concept study is to use functional magnetic resonance imaging and behavioral assessments to investigate the effect of citalopram on restricted repetitive behaviors in people with autism spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory status (outpatient) at time of consent
* Age 10-55 years
* Clinical diagnosis of Autism Spectrum Disorder
* IQ greater than or equal to 70
* Score greater than 8 on Children's Yale-Brown Obsessive Compulsive Scale
* Free of psychoactive medication for at least: one month for fluoxetine; two weeks for other SSRIs and neuroleptics; and five days for stimulants prior to MRI scanning [excepting stable doses (greater than three months duration) of anticonvulsant medication for seizure disorder]

Exclusion Criteria:

* Age less than 10 years or greater than 55 years, at time of consent
* Estimated IQ < 70
* Uncontrolled epilepsy (seizure within 6 months prior to consent)
* 4. Presence of medical conditions that might interfere with participation, or where participation would be contraindicated
* History of neurological injury: head trauma, poorly-controlled seizure disorder (seizure within the preceding six months), stroke, prior neurosurgery, or under the care of a neurologist or neurosurgeon as determined by interview
* History of claustrophobia
* Implanted or irremovable metal in the body (including certain tattoos and permanent make-up)
* Current pregnancy (as verified by testing prior to both initial dose administration of citalopram or placebo and prior to magnetic resonance imaging) due to the risk that may be associated with SSRI treatment and magnetic resonance imaging on fetal health
* Medical contraindications to SSRI therapy as determined by history (including induction of mania or hypomania during SSRI therapy, or known drug allergy)
* Concomitant medication that would interfere with study participation
* Prior history of citalopram treatment failure at appropriate doses and duration
* Prior history of treatment failure to two previous SSRI trials at appropriate doses and duration
* Ongoing need for psychoactive medication other than study medication [excepting stable doses (greater than three months duration) of anticonvulsant medication for seizure disorder, or diphenhydramine (Benadryl®)for sleep]

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging | two 2-hr scans
Clinicians Global Improvement Scale | Upon study completion

SECONDARY OUTCOMES:
Childrens Yale-Brown Obsessive Compulsive Scale | Baseline, wks 2, 4, 8, endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel S Dichter, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States